CLINICAL TRIAL: NCT01982994
Title: Intervention to Motivate Standing &Walking in Gastrointestinal Cancer Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, Niraj J. Gusani MD, Professor of Surgery and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 41440
Record Dates: First submitted 2013-10-28; First posted 2013-11-13 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Gastrointestinal Neoplasms
Keywords: Physical Activity Education; Caregivers
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education/Daily Planning (Experimental): Physical Activity Education and Daily Planning Tool
  Interventions: Behavioral: Education/Daily Planning
- No Education/Daily Planning (No Intervention): No Physical Activity Education/ Daily Planning Tool

INTERVENTIONS:
Behavioral: Education/Daily Planning — In this study, we will use educational materials delivered at the initial enrollment session and in daily "facts of the day" presented electronically to heighten awareness of (1) the risks of insufficient physical activity and excessive sedentary behavior, and (2) the expected beneficial outcomes of increased physical activity and reduced sedentary behavior. These messages should are designed to increase intentions to engage in physical activity and to limit sedentary behavior (motivational phase)
  Arms: Education/Daily Planning

SUMMARY:
Observational research has linked physical activity with faster recovery, improved quality of life, and greater survival; however, little is known about the effects of physical activity in pre-operative, peri-operative, or post-operative treatment contexts and there is a need for interventions to improve patient outcomes across the cancer treatment continuum. Three propositions derived from basic research, epidemiological evidence, and clinical practice informed our intervention development efforts: (1) Patient outcomes will be enhanced by interventions that increase physical activity (i.e., standing, walking) across the cancer treatment continuum (i.e., pre-operative, peri-operative, post-operative). (2) Reducing sedentary behavior (i.e., seated or reclined activities involving minimal energy expenditure) will enhance patient outcomes both by increasing physical activity and by stimulating additional adaptive physiological responses to reduced sedentary time (responses which are independent of physical activity-induced responses). (3) Patients with gastrointestinal cancers often suffer functional limitations that limit their independence and their health behaviors are strongly influenced by the family environment so interventions that engage caregivers (e.g., spouses) will be more effective than those that target patients/survivors alone.

DETAILED DESCRIPTION:
Phase 1 Screening and Baseline Assessment in Clinic Patients will be recruited by their physician upon diagnosis and immediately after the Penn State Surgical Oncology team presents then with the surgical treatment option. The patient must be able to identify an adult caregiver. The caregiver must be someone who is willing to participate in the study for the intervention period.

Once enrolled by the research assistant, the participant will complete an intake questionnaire to capture demographic information. The participant will then be given a tablet computer, training on how to use it to complete the questionnaires at the beginning and end of each day, an activity monitor with materials for securing it, and training on how/where to affix it on the leg.

In this study, we will use educational materials delivered at the initial enrollment session and in daily "facts of the day" presented electronically to heighten awareness of (1) the risks of insufficient physical activity and excessive sedentary behavior, and (2) the expected beneficial outcomes of increased physical activity and reduced sedentary behavior. These messages should are designed to increase intentions to engage in physical activity and to limit sedentary behavior (motivational phase). Although intentions are necessary for behavior change, a recent review of experimental evidence indicates that they are not sufficient. In the volitional phase, people translate those intentions into action by developing actions plans that specify when/where/how they will act (e.g., after lunch I will go on a 30 min walk around my neighborhood) and coping plans that specify how they will overcome anticipated barriers to desired behavior (e.g., if it rains after lunch, I will go to the mall to walk for 30 min). Repeated planning of this nature is the basis for breaking existing behavioral habits and forming newer (and hopefully more adaptive) ones. We have already developed an electronic daily planning tool that can be used at the beginning of each day to form action and coping plans for the target behaviors in this intervention. In the first two months of this project, we will tailor this existing planning tool for the target population by drawing from existing and emerging research on strategies for and barriers to health behaviors among cancer patients.

The control group will not receive the educational or daily planning components of the motivational intervention. They will, however, engage in self-monitoring by virtue of wearing activity monitors and using tablet computers to provide self-report data on their physical activity and sedentary behavior.

After the patient's surgery while staying at the Penn State Hershey Medical Center, the study coordinator will provide the caregiver with behavioral goals to help the patient recover from his/her surgery, and additional information about how the caregiver can support the patient's behavior change efforts.

Phase 2: Intervention Period

For the duration of the study, participant will:

* Complete beginning-and end -of-day questionnaires on the tablet computer. The beginning of day questionnaire will evaluate the patient's intentions and plans for daily physical activity. The end of day questionnaire will evaluate actual physical activity completed daily as well as the patient's physical, emotional, and social well-being.
* Wear and activity monitor

For participants in the experimental group the research assistant will also:

* Deliver the educational intervention for patients and caregivers during their first visit after they have signed the consent forms.
* Train patients how to use the daily planning tool prior to the beginning -of- day prior to the beginning-of-day questionnaires.

The theoretical basis for our intervention draws from both social-cognitive theory (i.e., Health Action Process Approach [HAPA]) and self-determination theory. The Health Action Process Approach differentiates between motivational and volitional phases of action control. In the motivational phase, people form intentions or goals for their behavior based on factors such as risk awareness and outcome expectations. In this study, we will use educational materials delivered at the initial enrollment session and in daily "facts of the day" presented electronically to heighten awareness of (1) the risks of insufficient physical activity and excessive sedentary behavior, and (2) the expected beneficial outcomes of increased physical activity and reduced sedentary behavior. These messages should are designed to increase intentions to engage in physical activity and to limit sedentary behavior (motivational phase). Although intentions are necessary for behavior change, a recent review of experimental evidence indicates that they are not sufficient. In the volitional phase, people translate those intentions into action by developing actions plans that specify when/where/how they will act (e.g., after lunch I will go on a 30 min walk around my neighborhood) and coping plans that specify how they will overcome anticipated barriers to desired behavior (e.g., if it rains after lunch, I will go to the mall to walk for 30 min). Repeated planning of this nature is the basis for breaking existing behavioral habits and forming newer (and hopefully more adaptive) ones. We have already developed an electronic daily planning tool that can be used at the beginning of each day to form action and coping plans for the target behaviors in this intervention. In the first two months of this project, we will tailor this existing planning tool for the target population by drawing from existing and emerging research on strategies for and barriers to health behaviors among cancer patients.

Self-determination theory posits that social factors, such as family relationships, can also influence motivation. Our recent work using experience sampling methodology and accelerometry has shown that spouses' autonomy support for patient physical activity and the spouse's level of physical activity were associated with patients' greater daily moderate physical activity and steps taken Individuals whose family members or health care providers show autonomy support for increasing physical activity and decreasing sedentary behavior are more likely to make those changes for reasons that come from within themselves and are freely chosen. Because close family members influence the emotional and physical well-being of patients, their inclusion in behavioral interventions is logical and has the potential to boost the effects of those interventions. In this study, caregivers will be educated about the importance of autonomy support in behavior change and strategies for supporting their partner's autonomy around physical activity and sedentary behavior change across the stages of treatment. This education will be delivered by the nurse coordinator at the initial education session following enrollment.

Collectively, these three components of patient education, daily planning, and caregiver education were assembled to strengthen intentions for desired health behaviors (motivational phase of behavior change), to increase the likelihood that such intentions will translate into action (volitional phase of behavior change), and to provide social resources that support behavior change in both of those phases.

The control group will not receive the educational or daily planning components of the motivational intervention. They will, however, engage in self-monitoring by virtue of wearing activity monitors and using tablet computers to provide self-report data on their physical activity and sedentary behavior.

During the intervention period the study coordinator will also contact the patient via phone weekly to ask questions related to the patients safety including questions about frequency of falls mild/moderate/severe, chest pain, dizziness, musculoskeletal soreness or pain, and changes in swelling.

Phase 3: Follow-Up Telephone Call

The research assistant will call the participant 30, 60, and 90 days after surgery to assess the frequency of hospital readmission or emergency room visits since being discharged.

Phase 4: Follow- Up Questionnaire

21 days after discharge form the hospital, participants and caregivers will complete a brief questionnaire that we will mail to them with a self-addressed stamped envelope.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gastrointestinal tract cancer (hepatobiliary) requiring surgical resection. for treatment
* Failing to meet the aerobic component of national physical activity guidelines over past week (e.g., < 150 min moderate-intensity physical activity or < 75 min vigorous-intensity physical activity).
* Excessive sedentary behavior over the past week (> 8 hrs/day sitting).
* Minimum age 18 years.
* A spouse or adult child serving as a caregiver who is also willing to participate.

Exclusion Criteria:

* Functional limitations that preclude normal physical activity.
* Patients who will be scheduled for surgery < 10 days after their clinic visit.
* Medical contraindications to physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with diagnosed gastrointestinal cancer who showed daily compliance using activity monitors and tablet computers to measure physical activity. | up to 1 year
  To demonstrate the feasibility and acceptability of using activity monitors and tablet computers to measure physical activity (standing, walking)/sedentary behavior (sitting) and deliver daily interventions in this patient population, we will evaluate daily compliance using activity monitors and tablet computers.

SECONDARY OUTCOMES:
Percentage of patients with a diagnosis of gastrointestinal cancer that benefit from an intervention of physical activity daily planning and education. | up to 1 year
  To evaluate the efficacy of this intervention, we will conduct a pilot study of a two-arm randomized controlled trial of the intervention against a self-monitoring control group.

CONTACTS AND LOCATIONS:
Overall Officials: Niraj J Gusani, M.D., M.S., Principal Investigator — Milton S. Hershey Medical Center; David E Conroy, Ph.D, Study Director — Penn State University
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Ballard-Barbash R, Friedenreich CM, Courneya KS, Siddiqi SM, McTiernan A, Alfano CM. Physical activity, biomarkers, and disease outcomes in cancer survivors: a systematic review. J Natl Cancer Inst. 2012 Jun 6;104(11):815-40. doi: 10.1093/jnci/djs207. Epub 2012 May 8. PMID 22570317
- [Background] Lynch BM. Sedentary behavior and cancer: a systematic review of the literature and proposed biological mechanisms. Cancer Epidemiol Biomarkers Prev. 2010 Nov;19(11):2691-709. doi: 10.1158/1055-9965.EPI-10-0815. Epub 2010 Sep 10. PMID 20833969
- [Background] Santos DA, Silva AM, Baptista F, Santos R, Vale S, Mota J, Sardinha LB. Sedentary behavior and physical activity are independently related to functional fitness in older adults. Exp Gerontol. 2012 Dec;47(12):908-12. doi: 10.1016/j.exger.2012.07.011. Epub 2012 Aug 1. PMID 22884978
- [Background] Carlson SA, Fulton JE, Schoenborn CA, Loustalot F. Trend and prevalence estimates based on the 2008 Physical Activity Guidelines for Americans. Am J Prev Med. 2010 Oct;39(4):305-13. doi: 10.1016/j.amepre.2010.06.006. PMID 20837280
- [Background] Matthews CE, Chen KY, Freedson PS, Buchowski MS, Beech BM, Pate RR, Troiano RP. Amount of time spent in sedentary behaviors in the United States, 2003-2004. Am J Epidemiol. 2008 Apr 1;167(7):875-81. doi: 10.1093/aje/kwm390. Epub 2008 Feb 25. PMID 18303006
- [Background] Schwarzer R, Lippke S, Luszczynska A. Mechanisms of health behavior change in persons with chronic illness or disability: the Health Action Process Approach (HAPA). Rehabil Psychol. 2011 Aug;56(3):161-70. doi: 10.1037/a0024509. PMID 21767036
- [Background] Gonzalez M, Guillaume JE, Laloux P, Mahieu P, Installe E. Strychnine poisoning, hypoxic damage, severe acidosis: a case report. Acta Clin Belg Suppl. 1990;13:94-5. No abstract available. PMID 2239073
- [Background] Martire LM, Stephens MA, Mogle J, Schulz R, Brach J, Keefe FJ. Daily spousal influence on physical activity in knee osteoarthritis. Ann Behav Med. 2013 Apr;45(2):213-23. doi: 10.1007/s12160-012-9442-x. PMID 23161472
- [Background] Martire LM, Schulz R, Helgeson VS, Small BJ, Saghafi EM. Review and meta-analysis of couple-oriented interventions for chronic illness. Ann Behav Med. 2010 Dec;40(3):325-42. doi: 10.1007/s12160-010-9216-2. PMID 20697859